CLINICAL TRIAL: NCT00137566
Title: The Effect of Paracetamol in the Treatment of Non-severe Malaria in Children in Guinea-Bissau
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Responsible Party: Poul-Erik Kofoed, Bandim Health Project
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSB-2004-paracetamol
Record Dates: First submitted 2005-08-28; First posted 2005-08-30 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Malaria; Falciparum
Keywords: malaria; treatment; paracetamol; chloroquine; Guinea-Bissau; children; P.falciparum
MeSH Terms: conditions — Malaria | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 Paracetamol (Experimental): Paracetamol as per protocol
  Interventions: Drug: acetaminophen (paracetamol)
- 2 Placebo (Placebo Comparator): Inactive placebo as per protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: acetaminophen (paracetamol) — Paracetamol tablets, 50 mg/kg/day for 3 days.
  Arms: 1 Paracetamol
Other: Placebo
  Arms: 2 Placebo

SUMMARY:
The National Malaria Programme in Guinea-Bissau recommends paracetamol for all children treated for malaria. We, the investigators of the Bandim Health Project, want to evaluate whether this treatment has any effect on:

* the well-being of the child;
* the parasite clearance time; and
* the rate of a re-appearance of parasites during 35 days of follow-up.

Children presenting at Bandim Health Centre with malaria will be treated with chloroquine plus paracetamol or chloroquine plus placebo. Blood samples will be obtained daily for the first 4 days and then once a week until day 35.

DETAILED DESCRIPTION:
A Cochrane Review was unable to show a superior antipyretic effect of paracetamol compared with placebo in febrile children. Recent research suggests that the time to parasite clearance in non-severe malaria is longer in children being given paracetamol. As the costs associated with the use of paracetamol is not trivial and the risk of adverse effects is not negligible, we want to evaluate the effects of paracetamol on:

* the well-being of the child;
* the parasite clearance time; and
* the recrudescence rate.

Children presenting at Bandim Health Centre with symptoms of malaria and a malaria film showing mono-infection with P.falciparum will, following consent to participate, randomly be allocated to treatment with chloroquine and paracetamol or with chloroquine and placebo.

Blood samples will be obtained daily for the first 4 days. The children will be visited and a malaria film taken on day 7 and then weekly until day 35. On inclusion and whenever parasitaemia is detected a capillary blood sample will be taken for PCR analyses to be able to distinguish re-infection from recrudescence.

During follow-up children are recommended to present at the health centre in case of persistent fever or any other symptoms. Examination and treatment will be free of charge. Whenever a child has re-infection sulfadoxine/pyrimethamine will be used for re-treatment following the recommendation of the National malaria Programme.

After the inclusion of 80 children a preliminary analysis will be performed. If 50% or more of the children in any of the study arms have reappearing parasitaemia the study will be terminated.

If the parasite clearance time and especially the recrudescence rate is higher for children being given paracetamol the current recommendation from the National Malaria Programme should be reconsidered. If children treated with paracetamol feel better during the acute illness making it more likely for them to have en adequate intake of food and liquid this benefit should be considered in the evaluation of the current recommendations.

ELIGIBILITY:
Inclusion Criteria:

* < 15 years of age
* Presenting at Bandim Health Centre
* Symptoms suggestive of malaria
* At least 20 P. falciparum parasites per 200 leukocytes
* Live in Bandim (to enable follow-up)

Exclusion Criteria:

* Severely ill children considered to need the services of a hospital by the doctor in charge
* Previous idiosyncratic reactions to chloroquine or paracetamol

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-05; Primary Completion 2006-11 (Actual); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
parasite clearance time | 35 days
recrudescence rate | 35 days

SECONDARY OUTCOMES:
well-being of the child | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Professor, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau Region, Guinea-Bissau

REFERENCES:
- [Background] Russell FM, Shann F, Curtis N, Mulholland K. Evidence on the use of paracetamol in febrile children. Bull World Health Organ. 2003;81(5):367-72. Epub 2003 Jul 7. PMID 12856055
- [Derived] Jovel IT, Kofoed PE, Rombo L, Rodrigues A, Ursing J. Temporal and seasonal changes of genetic polymorphisms associated with altered drug susceptibility to chloroquine, lumefantrine, and quinine in Guinea-Bissau between 2003 and 2012. Antimicrob Agents Chemother. 2015 Feb;59(2):872-9. doi: 10.1128/AAC.03554-14. Epub 2014 Nov 24. PMID 25421474
- [Derived] Kofoed PE, Ursing J, Rodrigues A, Rombo L. Paracetamol versus placebo in treatment of non-severe malaria in children in Guinea-Bissau: a randomized controlled trial. Malar J. 2011 Jun 1;10:148. doi: 10.1186/1475-2875-10-148. PMID 21631932